CLINICAL TRIAL: NCT04530981
Title: A Phase 1 Open-label, Multicenter Study to Evaluate the Effect of Ripretinib on the Pharmacokinetics of a CYP2C8 Probe Substrate (Repaglinide) in Patients with Advanced Gastrointestinal Stromal Tumors (GIST)
Brief Title: A Drug-Drug Interaction Study to Evaluate the Effect of Ripretinib on the Pharmacokinetics of a CYP2C8 Probe Substrate in Patients with Advanced GIST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2618-01-007
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: GIST - Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Repaglinide 0.5 mg + Ripretinib 150 mg QD (Experimental): A single dose of repaglinide 0.5 mg (1 × 0.5-mg tablet) will be administered orally on Cycle 1 Day 1 and Cycle 1 Day 15. Ripretinib 150 mg QD (3 × 50-mg tablets) will be administered orally from Day 2 through Day 28 for Cycle 1 and will be administered continuously from Cycle 2 until disease progression as assessed by the Investigator, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Ripretinib; Drug: Repaglinide

INTERVENTIONS:
Drug: Ripretinib — Oral KIT/PDGFRA kinase inhibitor
  Other Names: QINLOCK
Drug: Repaglinide — Oral antihyperglycemic agent

SUMMARY:
Evaluate the Effect of Ripretinib on the Pharmacokinetics of a CYP2C8 Substrate

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age.
2. Patients must have a histologic diagnosis of GIST.
3. Patients must have GIST that has progressed on or have intolerance to at least 2 lines of prior TKI therapies.
4. Patients must have an Eastern Cooperative Oncology Group performance score of ≤ 2.
5. If a female of childbearing potential, must have a negative pregnancy test prior to enrollment and agree to follow the contraception requirements.
6. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Received prior anticancer or other investigational therapy within 28 days or 5× the half-life prior to the first dose.
2. Prior treatment with ripretinib.
3. Patients who have had prior repaglinide treatment within 14 days prior to Cycle 1 Day 1.
4. History or presence of clinically relevant cardiovascular abnormalities.
5. Gastrointestinal abnormalities including but not limited to:

   * inability to take oral medication,
   * malabsorption syndromes,
   * requirement for intravenous alimentation.
6. Patients who have type 1 or type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration for Repaglinide | Cycle 1 Day 1 and Cycle 1 Day 15 (pre-dose and at multiple time points [up to 24 hours] post-dose). Each cycle is 28 days.
  Measure the Cmax
Area under the concentration-time curve (AUC) from time 0 up to time t (AUC0-t) for Repaglinide | Cycle 1 Day 1 and Cycle 1 Day 15 (pre-dose and at multiple time points [up to 24 hours] post-dose). Each cycle is 28 days.
  Measure the AUC0-t
AUC from time 0 and extrapolated to infinity (AUC0-∞) | Cycle 1 Day 1 and Cycle 1 Day 15 (pre-dose and at multiple time points [up to 24 hours] post-dose). Each cycle is 28 days.
  Measure the AUC0-∞

SECONDARY OUTCOMES:
Incidence of Adverse Events | Cycle 1 through study completion (~ 12 months). Each cycle is 28 days.
  Adverse events [TEAEs, SAEs], dose reduction, dose interruption, or discontinuation, vital signs (heart rate [beats/min], and changes in laboratory parameters (chemistry, hematology, urinalysis, coagulation).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No